CLINICAL TRIAL: NCT02010567
Title: Phase Ib/II Study of Neoadjuvant Chemoradiotherapy With CRLX-101 and Capecitabine for Locally Advanced Rectal Cancer
Brief Title: Neoadjuvant Chemoradiotherapy With CRLX-101 and Capecitabine for Rectal Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The study was halted prematurely at the funding partner's request.
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: Cerulean Pharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC 1315
Record Dates: First submitted 2013-12-09; First posted 2013-12-12 (Estimated); Results first posted 2017-11-14 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-10

CONDITIONS: Rectal Cancer
Keywords: rectal cancer; colorectal cancer; locally advanced rectal cancer; locally advanced rectal cancer (resectable); locally advanced rectal cancer (non-resectable); chemoradiotherapy; nanopharmaceutical; CLRX101; camptothecin; capecitabine
MeSH Terms: conditions — Rectal Neoplasms; Colorectal Neoplasms | interventions — IT-101; Capecitabine; Radiotherapy; Radiotherapy, Intensity-Modulated; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CLRX101 MTD/RP2D (Experimental): During Phase Ib, we will evaluate the safety and determine the MTD/RP2D of CRLX101 + capecitabine (Cape) and radiation therapy (XRT) in patients with rectal cancer using the traditional 3+3 dose escalation design. Adverse events (AEs) will be evaluated via the CTCAE version 4.0. Patients in Phase Ib will also be followed for pathological response if they have resectable disease.
  Interventions: Drug: CRLX101; Drug: Capecitabine; Radiation: Radiotherapy
- Chemoradiotherapy + Surgery (Experimental): In Phase II, CRLX101 will be administered at the RP2D in combination with capecitabine and radiation in patients with locally advanced rectal cancer for a total of 5-6 weeks, depending on the total radiation dose. A total of 3 doses of CRLX101 will be administered every other week. Surgery will take place at least 6 weeks after the completion of chemoradiotherapy.
  Interventions: Drug: CRLX101; Drug: Capecitabine; Radiation: Radiotherapy; Procedure: Surgery

INTERVENTIONS:
Drug: CRLX101 — CRLX101 is an experimental nanoparticle formulation of the anticancer agent camptothecin manufactured by Cerulean Pharma Inc..
Drug: Capecitabine — Capecitabine is an oral fluoropyrimidine pro-drug, metabolically converted to 5-fluorouracil after administration. It is indicated as adjuvant treatment in patients with stage III colorectal cancer (Dukes' C colon cancer), and as first-line treatment of metastatic colorectal cancer.
  Other Names: Xeloda
Radiation: Radiotherapy — This protocol allows physician discretion as to the use of Intensity Modulated Radiation Therapy (IMRT) or 3D conformal planning techniques.
  Radiation begins on Day1 of neoadjuvant chemotherapy and continues for 28 (if <T4) or 30 (T4 disease) consecutive weekdays. Patient will receive 1.8 Gy daily fractions of radiotherapy without a break except for weekends and holidays.
  Dose is to be prescribed to an isodose surface that encompasses the planning target volume (PTV) and that satisfies the dose uniformity guidelines below. The minimum dose to PTV 1 and PTV 2 shall be no less than 95% of the protocol specified dose for that volume.
  Other Names: Intensity Modulated Radiation Therapy; IMRT
Procedure: Surgery — Surgery will take place at least 6 weeks post completion of chemoradiotherapy in patients with resectable disease; tissue from surgical resection will be preserved for correlative studies in those patients who do not achieve a pCR.
  Other Names: Resection; Surgical resection
  Arms: Chemoradiotherapy + Surgery

SUMMARY:
This trial will enroll patients with locally advanced rectal cancer (resectable and non-resectable).The phase Ib dose escalation portion of trial is designed to determine the maximum tolerated dose (MTD) of CRLX101 when combined with standard neoadjuvant therapies capecitabine (Cape) and radiation therapy (XRT). CRLX101 is a nanopharmaceutical (NP) formulation of camptothecin. These results will determine the recommended phase II dose (RP2D) for CRLX101 in this setting. The phase II portion of the trial is designed to evaluate the efficacy and safety of CRLX101 at the RP2D, when combined with capecitabine and radiation therapy prior to surgery.

DETAILED DESCRIPTION:
This is an open label, single-arm, multi-center, Phase Ib/II study designed to evaluate CRLX101, which is a NP formulation of camptothecin, dosed in combination with capecitabine and radiation therapy in patients with advanced rectal carcinoma.

The purpose of the Phase Ib portion of this study is to identify the MTD of CRLX101 when added to standard neoadjuvant chemo-radiotherapy. The MTD will be based on the rate of dose-limiting toxicity (DLT) in Phase Ib, and will be assessed via NCI's CTCAE v4.0 toxicity criteria. The MTD will be assigned as the RP2D in this trial.

If CRLX101 can be safely administered in combination with capecitabine and radiation at doses >/= 9 mg/m^2 IV in the Phase Ib study, then the trial will proceed to Phase II. Patients in the Phase Ib study will be included in the Phase II outcome analyses when applicable. The phase II study is designed to evaluate the efficacy of this regimen by assessing the rate of pathological complete response (pCR) while monitoring safety and tolerability.

We anticipate accrual of up to 25 patients per year for the Phase II study, with a slightly faster accrual of 2-3 patients per month for Phase Ib given the broader inclusion criteria.

During Phase Ib, we will evaluate the safety and determine the MTD/RP2D of CRLX101 + capecitabine (Cape) and radiation therapy (XRT) in patients with rectal cancer using the traditional 3+3 dose escalation design. Adverse events (AEs) will be evaluated via the CTCAE version 4.0. Patients in Phase Ib will also be followed for pathological response if they have resectable disease.

If CRLX101 can be safely administered in combination with capecitabine and radiation at doses >/=9 mg/m^2 IV in the Phase Ib study, then the trial will proceed to Phase II with a primary objective of estimating the rate of pCR. Non-metastatic patients with resectable disease and treated at the MTD/RP2D in Phase Ib will be included in the Phase II study population.

In Phase II, CRLX101 will be administered at the RP2D in combination with capecitabine and radiation in patients with locally advanced rectal cancer for a total of 5-6 weeks, depending on the total radiation dose. A total of 3 doses of CRLX101 will be administered every other week. Surgery will take place at least 6 weeks after the completion of chemoradiotherapy.

For our non-metastatic Phase I patients and our Phase II population, postoperative adjuvant therapy is indicated regardless of whether a pCR is achieved or not. While there are a number of regimens used in the adjuvant setting, national guidelines do not specify one of these regimens over the other. Given the consistent application of adjuvant therapies in this population, we also plan to follow Phase II patients for both disease free survival (DFS) and overall survival (OS).

ELIGIBILITY:
Inclusion Criteria:

1. Eastern Cooperative Oncology Group (ECOG) performance score ≤ 2
2. Phase Ib and II: surgical candidates, with moderate to high-risk pathologically-confirmed rectal cancer (Tumor (T) and Nodal (N) stage cT3-4N0 or cT1-4N+); clinical staging by endoscopic ultrasound (EUS) or magnetic resonance imaging (MRI) is permitted.

   Phase Ib only:
   * Patients with metastatic rectal cancer are allowed if their primary site meets other eligibility criteria and chemoradiotherapy is recommended as initial therapy for symptom palliation by the multidisciplinary treating team
   * Patients with locally advanced unresectable rectal cancer are allow provided:

     * There is no evidence of recto-vaginal, recto-vesicular, recto-intestinal fistulization
     * Standard dose and schedule chemoradiotherapy is recommended as initial therapy by the multidisciplinary treating team
3. Age ≥18 years old
4. Women of childbearing potential (WOCBP) must have negative pregnancy test within 7 days prior to D1 of treatment
5. Recommendation to undergo concurrent chemoradiation, as determined by the treating physician
6. Ability to swallow oral medications
7. As determined by the enrolling physician or protocol designee, ability of the patient to understand and comply with study procedures for the entire length of the study
8. Informed consent reviewed and signed

Exclusion Criteria:

Patients meeting any of the following exclusion criteria will not be able to participate in this study:

1. Grade 2 or higher diarrhea at baseline unless deemed by the investigator to be caused by laxatives prescribed for symptomatic partial obstruction (e.g. MiraLAX®)
2. Not deemed a candidate for concurrent chemoradiation for medical reasons, such as uncontrolled infection (including HIV), uncontrolled diabetes mellitus or cardiac disease which, in the opinion of the treating physician, would make this protocol unreasonably hazardous for the patient.
3. Specific laboratory exclusion values, including:

   * Hemoglobin < 10.0 g/dL for males and ≤ 9.0 g/dL for females (transfusion allowed to achieve or maintain levels)
   * Absolute neutrophil count (ANC) < 1,500/mm3
   * Platelet count < 100,000/mm3
   * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) > 2.5 times upper level of normal (ULN)
   * Alkaline phosphatase > 2.5 times ULN
   * Total bilirubin > 1.5 times ULN
   * Creatinine clearance < 50 mL/min
   * International normalized ratio (INR) >2
4. Known dihydropyrimidine dehydrogenase (DPD) deficiency
5. History of Gilbert's syndrome
6. Those who require therapeutic anticoagulation with coumarin-derivative anticoagulants
7. Unable to provide informed consent
8. Receiving any other concurrent cytotoxic, biologic agent(s) or investigational agent
9. Patients with a "currently active" second malignancy other than non-melanoma skin cancers, non-invasive bladder cancer, "low risk" adenocarcinoma of the prostate and carcinoma in situ of the cervix. Patients are not considered to have a "currently active" malignancy if they have completed therapy and are free of disease for ≥ 2 years.
10. Previous pelvic radiation therapy
11. Prior treatment with a topoisomerase I inhibitor (i.e. irinotecan, topotecan)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2013-12; Primary Completion 2016-09-16 (Actual); Study Completion 2019-06-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Wang, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (6):
- United States (6):
  - Rocky Mountain Cancer Center, Denver, Colorado
  - Indiana University Simon Cancer Center, Indianapolis, Indiana
  - University of North Carolina, Chapel Hill, North Carolina
  - Rex Cancer Center at Rex Hospital, Raleigh, North Carolina
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Swedish Cancer Institute, Seattle, Washington

REFERENCES:
- [Derived] Sanoff HK, Moon DH, Moore DT, Boles J, Bui C, Blackstock W, O'Neil BH, Subramaniam S, McRee AJ, Carlson C, Lee MS, Tepper JE, Wang AZ. Phase I/II trial of nano-camptothecin CRLX101 with capecitabine and radiotherapy as neoadjuvant treatment for locally advanced rectal cancer. Nanomedicine. 2019 Jun;18:189-195. doi: 10.1016/j.nano.2019.02.021. Epub 2019 Mar 8. PMID 30858085
- [Derived] Tian X, Nguyen M, Foote HP, Caster JM, Roche KC, Peters CG, Wu P, Jayaraman L, Garmey EG, Tepper JE, Eliasof S, Wang AZ. CRLX101, a Nanoparticle-Drug Conjugate Containing Camptothecin, Improves Rectal Cancer Chemoradiotherapy by Inhibiting DNA Repair and HIF1alpha. Cancer Res. 2017 Jan 1;77(1):112-122. doi: 10.1158/0008-5472.CAN-15-2951. Epub 2016 Oct 26. PMID 27784746
- See also: Lineberger Comprehensive Cancer Center website — http://unclineberger.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from 5 medical institutions between December 2013 and September 2016
Pre-assignment Details: A total of 39 patients were consented to this study; 4 patients were found ineligible, 3 withdrew prior to treatment, leaving 32 patients who went on study.
Groups:
- Cohort A, Phase Ib, Dose Level 1: CRLX101 12mg/ m^2 , via intravenous catheter (IV), on Monday, every other week for the first five weeks of chemoradiation.
  Capecitabine 825mg/ m^2 PO BID, M-F XRT 180 cGy/day, M-F for 6 weeks
- Cohort A, Phase Ib, Dose Level 2; Cohort A, Phase II, Dose Level 2: CRLX101 15mg/ m^2 , via intravenous catheter (IV), on Monday, every other week for the first five weeks of chemoradiation.
  Capecitabine 825mg/ m^2 PO BID, M-F XRT 180 cGy/day, M-F for 6 weeks
- Cohort B, Phase Ib, Dose Level 1, Weekly: CRLX101 12mg/ m^2 , via intravenous catheter (IV), on Monday, every week for the first five weeks of chemoradiation.
  Capecitabine 825mg/ m^2 PO BID, M-F XRT 180 cGy/day, M-F for 6 weeks
- Cohort B, Phase Ib, Dose Level 2, Weekly: CRLX101 15mg/ m^2 , via intravenous catheter (IV), on Monday, every week for the first five weeks of chemoradiation.
  Capecitabine 825mg/ m^2 PO BID, M-F XRT 180 cGy/day, M-F for 6 weeks
Period: Overall Study
Arm/Group | Cohort A, Phase Ib, Dose Level 1 | Cohort A, Phase Ib, Dose Level 2 | Cohort A, Phase II, Dose Level 2 | Cohort B, Phase Ib, Dose Level 1, Weekly | Cohort B, Phase Ib, Dose Level 2, Weekly
Started | 3 | 6 | 14 | 3 | 6
Completed | 3 | 6 | 13 | 3 | 5
Not Completed | 0 | 0 | 1 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Cohort A, Phase Ib, Dose Level 1: CRLX101 12mg/ m^2 , via intravenous catheter (IV), on Monday, every other week for the first five weeks of chemoradiation.
  Capecitabine 825mg/ m^2 by mouth two times a day (PO BID), Monday through Friday (M-F) XRT 180 centigray (cGy)/day, M-F for 6 weeks
- Total: Total of all reporting groups
Arm/Group | Cohort A, Phase Ib, Dose Level 1 | Cohort A, Phase Ib, Dose Level 2 | Cohort A, Phase II, Dose Level 2 | Cohort B, Phase Ib, Dose Level 1, Weekly | Cohort B, Phase Ib, Dose Level 2, Weekly | Total
Number analyzed (Participants) | 3 | 6 | 14 | 3 | 6 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 4 | 14 | 3 | 5 | 28
  >=65 years | 1 | 2 | 0 | 0 | 1 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 4 | 0 | 3 | 10
  Male | 1 | 5 | 10 | 3 | 3 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 3 | 0 | 1 | 5
  White | 3 | 5 | 11 | 3 | 4 | 26
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 6 | 14 | 3 | 6 | 32

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of CRLX101 When Added to Standard Neoadjuvant Chemoradiotherapy Consisting of Capecitabine + Radiotherapy in Locally Advanced Rectal Cancer
Description: The MTD is the highest dose of CRLX101 at which ≤1 out of 6 patients had a dose limiting toxicity (DLT) using CTCAE v4.0 toxicity criteria. DLTs include Grade (G) >3 neutropenia for ≥7 days; G 3 or 4 neutropenia with fever; G 4 anemia not related to cancer-associated bleeding; G 4 thrombocytopenia or G 3 with clinically significant bleeding; G ≥3 nausea or vomiting >48 hours despite anti-emetics; G 2 cystitis not resolved within 14 days; second G 2 cystitis; G 3 or 4 cystitis; diarrhea requiring dose reduction; Any other non-hematologic toxicity G ≥3 requiring a dose reduction (G ≥3 infusion-related reactions were not a DLT unless they recur despite slowing down the infusion); Other CRLX101 related treatment emergent adverse effect (TEAE) that requires patient withdrawal prior to completing all doses; Radiotherapy interruption due to TEAEs ≥5 days; or Dose interruption or reduction of capecitabine due to TEAE that results in <50% of the scheduled capecitabine dose for entire course
Time Frame: 12 weeks
Population: Since this objective applies only to Phase Ib patients, the Phase II cohort patients were not included
Measure: Number; unit: mg/m^2 every other week
Groups:
- Dose Escalation Phase Ib: Phase Ib patients who received at least one dose of CRLX101 at either 12mg/m2 or 15mg/m2 either every other week (Cohort A) or weekly (Cohort B)
Arm/Group | Dose Escalation Phase Ib
Number analyzed (Participants) | 18
mg/m^2 every other week | 15

2. Primary Outcome: Pathological Complete Response (pCR) Rate
Description: Primary Objective Phase II: Pathological response will be made based on microscopic assessment of the surgical specimen at the primary treatment site. A pCR must include no gross or microscopic tumor identified anywhere within the surgical specimen. This must include:No evidence of malignant cells in the primary tumor specimen and No lymph nodes that contain tumor.
Time Frame: 12 weeks
Measure: Number (95% Confidence Interval); unit: percentage of participants with pCR
Groups:
- All Participants: All resectable participants who received CRLX101 + capecitabine (Cape) and radiation therapy (XRT) regardless of dose and timing of treatment
Arm/Group | All Participants
Number analyzed (Participants) | 32
percentage of participants with pCR | 19 [7 to 36]

3. Secondary Outcome: Pathological Response Rate
Description: Pathologic response will be made based on microscopic assessment of the surgical specimen at the primary treatment site, including regional nodes and any peritumoral satellite nodules in the specimen, and categorized as outlined below as per the American Joint Committee on Cancer (AJCC) Cancer Staging Manual 7th edition.Determination of pathological response will be reported by the local pathologist.
  * Pathologic Complete Response (pCR): No gross or microscopic tumor identified anywhere within the surgical specimen. This must include: No evidence of malignant cells in the primary tumor specimen and No lymph nodes that contain tumor.
  * Moderate response: Single cells or small groups of cancer cells
  * Minimal response: Residual cancer outgrown by fibrosis
  * Poor response:Minimal or no tumor kill; extensive residual cancer
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 32
Participants
  pCR | 6
  Moderate response | 18
  Minimal response | 7
  Unknown | 1

4. Secondary Outcome: Number of Participants With Grade 3 or Higher, Treatment-related Toxicities
Description: Toxicity profile of CRLX101 when combined with capecitabine + radiotherapy to treat patients with locally advanced rectal cancer. Phase Ib and Phase II - Safety is the reported adverse event (AE) profile characterized by NCI CTCAE v4.0. The profile was limited to grade 3 or higher, treatment related AEs.
Time Frame: 12 weeks
Measure: Number; unit: participants with AE
Arm/Group | All Participants
Number analyzed (Participants) | 32
participants with AE
  Colitis | 1
  Dermatitis, radiation | 1
  Diarrhea | 1
  Hypophosphatemia | 1
  Lymphocyte count decreased | 9
  Rectal obstruction | 1
  White blood cell decreased | 1

5. Secondary Outcome: Disease-free Survival (DFS) Rate
Description: Phase II only - DFS will be defined as the time from surgical resection until disease recurrence or death as a result of any cause, reported as the count of participants still alive without recurrence at the end of study follow-up.
Time Frame: An average of 2.6 years (full range 2.1 to 3.1 years)
Population: 14 of 32 participants were enrolled in the Phase II portion of the study. Of these 14, one participant withdrew prior to surgery and was therefore not evaluable for this outcome
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A, Phase II, Dose Level 2
Number analyzed (Participants) | 13
Participants | 10

6. Secondary Outcome: Overall Survival (OS) Rate
Description: Phase II only - OS is defined as the time from surgical resection until death reported as the count of participants still alive at the end of study follow-up.
Time Frame: an average of 2.6 years (full range 2.1 to 3.1 years)
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A, Phase II, Dose Level 2
Number analyzed (Participants) | 13
Participants | 13

7. Secondary Outcome: Disease-free Survival (DFS) Rate Based on Pathological Complete Response (pCR).
Description: Phase II only - a comparison of DFS for patients who achieve pCR and those who do not. DFS will be defined as the time from surgical resection until disease recurrence or death as a result of any cause, reported as the count of participants still alive without recurrence at the end of study follow-up.
Time Frame: an average of 2.6 years (full range 2.1 to 3.1 years)
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A, Phase II, Dose Level 2
Number analyzed (Participants) | 13
Participants
  pathological complete response (pCR): number analyzed (Participants) | 2
  pathological complete response (pCR) | 2
  Did not achieve pCR: number analyzed (Participants) | 11
  Did not achieve pCR | 8

8. Secondary Outcome: Overall Survival (OS) Based on Pathological Complete Response (pCR).
Description: Phase II only - a comparison of OS for patients who achieve pCR and those who do not. OS is defined as the time from surgical resection until death reported as the count of participants still alive at the end of study follow-up.
Time Frame: an average of 2.6 years (full range 2.1 to 3.1 years)
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A, Phase II, Dose Level 2
Number analyzed (Participants) | 13
Participants
  pathological complete response (pCR): number analyzed (Participants) | 2
  pathological complete response (pCR) | 2
  Did not achieve pCR: number analyzed (Participants) | 11
  Did not achieve pCR | 11

ADVERSE EVENTS:
Time Frame: Adverse events were collected up to 30 days after treatment was discontinued (approximately 12 weeks from study entry)
Description: All patients were evaluated for serious adverse events (SAEs)
Groups:
- Cohort A, Phase Ib, Level 1: 12mg/m^2 CRLX101 every other week + 825mg/m^2 BID Capecitabine + XRT
- Cohort A, Phase Ib, Level 2: 15mg/m^2 CRLX101 every other week + 825mg/m^2 BID Capecitabine + XRT
- Cohort A, Phase II, Level 2; Cohort B, Phase Ib, Level 2: 15mg/m^2 CRLX101 IV weekly + 825mg/m^2 BID Capecitabine + XRT
- Cohort B, Phase Ib, Level 1: 12mg/m^2 CRLX101 IV weekly + 825mg/m^2 BID Capecitabine + XRT
Arm/Group | Cohort A, Phase Ib, Level 1 | Cohort A, Phase Ib, Level 2 | Cohort A, Phase II, Level 2 | Cohort B, Phase Ib, Level 1 | Cohort B, Phase Ib, Level 2
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/6 | 0/14 | 0/3 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/6 | 1/14 | 0/3 | 0/6
Other Adverse Events (participants affected / at risk) | 3/3 | 6/6 | 14/14 | 3/3 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A, Phase Ib, Level 1 (N=3) | Cohort A, Phase Ib, Level 2 (N=6) | Cohort A, Phase II, Level 2 (N=14) | Cohort B, Phase Ib, Level 1 (N=3) | Cohort B, Phase Ib, Level 2 (N=6)
Colonic obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A, Phase Ib, Level 1 (N=3) | Cohort A, Phase Ib, Level 2 (N=6) | Cohort A, Phase II, Level 2 (N=14) | Cohort B, Phase Ib, Level 1 (N=3) | Cohort B, Phase Ib, Level 2 (N=6)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 4 (4) | 2 (2) | 0 (0) | 3 (3)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Anal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 4 (4) | 11 (11) | 2 (2) | 4 (4)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 4 (4) | 1 (1) | 2 (2)
Anxiety (Psychiatric disorders) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Bladder spasm (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bloating (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholesterol high (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 4 (4) | 4 (4) | 3 (3) | 1 (1)
Creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cystitis noninfective (Renal and urinary disorders) | 0 (0) | 2 (2) | 4 (4) | 1 (1) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis radiation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 4 (4) | 10 (10) | 0 (0) | 5 (5)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Edema limbs (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 2 (2) | 3 (3) | 11 (11) | 2 (2) | 5 (5)
Fever (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Hemorrhoids (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 4 (4) | 5 (5) | 0 (0) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 2 (2)
Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 5 (5) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 0 (0) | 3 (3) | 4 (4) | 1 (1) | 1 (1)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 3 (3) | 2 (2) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (3) | 3 (3) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 4 (4)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 4 (4) | 3 (3) | 3 (3)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infusion related reaction (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 3 (3) | 3 (3) | 8 (8) | 2 (2) | 4 (4)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 3 (3) | 5 (5) | 1 (1) | 2 (2)
Neutrophil count decreased (Investigations) | 2 (2) | 0 (0) | 2 (2) | 2 (2) | 3 (3)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Perineal pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 3 (3) | 3 (3) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1) | 2 (2) | 5 (5) | 1 (1) | 1 (1)
Rectal mucositis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rectal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal pain (Gastrointestinal disorders) | 3 (3) | 3 (3) | 4 (4) | 3 (3) | 3 (3)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 1 (1) | 2 (2) | 5 (5) | 2 (2) | 2 (2)
Urinary tract pain (Renal and urinary disorders) | 3 (3) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Urinary urgency (Renal and urinary disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Vaginal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Vaginal pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Weight loss (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
White blood cell decreased (Investigations) | 3 (3) | 2 (2) | 5 (5) | 2 (2) | 3 (3)

LIMITATIONS AND CAVEATS:
Follow-up of participants was ended early, resulting in few or no observed events (progression or death) for all survival endpoints.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes